CLINICAL TRIAL: NCT00473434
Title: An Open Label Multicentre Study to Determine the Dose Distribution of Paliperidone ER in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013213; R076477SCH3021
Record Dates: First submitted 2007-05-11; First posted 2007-05-15 (Estimated); Results first posted 2012-10-08 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Drug Therapy; Treatment Outcome
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Experimental): Paliperidone3mg or 6mg or 9mg or 12mg once daily for 52 weeks
  Interventions: Drug: Paliperidone

INTERVENTIONS:
Drug: Paliperidone — 3mg or 6mg or 9mg or 12mg once daily for 52 weeks

SUMMARY:
The purpose of this trial is to evaluate the dose distribution, effectiveness and safety in patients with schizophrenia who are switched from an oral atypical antipsychotic to Paliperidone ER. In this study patients and physicians know the name and the dose of the study drug. Newly diagnosed patients will also be included in the study. In general, the recommended Paliperidone ER dose will be 6 mg once daily, however some patients may require a higher or lower initial dose in the recommended range of 3 to 12 mg once daily. The dose can be adjusted any point during the study, to a maximum dose of 12mg/day. Flexible dosing was chosen to best mimic actual clinical practice.The safety assessments to be conducted throughout this study including the regular monitoring and recording of all Adverse Events and Serious Adverse Events.

DETAILED DESCRIPTION:
This trial is a non-randomised (both patient and physician know the study drug), single arm, open label multicentre study which is aimed to evaluate the dose distribution, efficacy and safety in patients with schizophrenia who are switched from an oral atypical antipsychotic to Paliperidone ER. Newly diagnosed patients will also be included in the study. In general, the recommended Paliperidone ER dose will be 6 mg once daily, however some patients may require a higher or lower initial dose in the recommended range of 3 to 12 mg once daily. The dose can be adjusted any point during the study, to a maximum dose of 12mg/day. Flexible dosing was chosen to best mimic actual clinical practice.The study duration will be split into two phases. Phase A will be 12 weeks and Phase B which will be an optional follow up phase will be 40 weeks. Assessment of efficacy and safety will be performed in Phase A at baseline, 2, 4, 6, 9 and 12 weeks and in Phase B at 20, 28, 36, 44 and 52 weeks. At the first visit, a full psychiatric history, demographic data and physical examination will be undertaken. Throughout the study, the following procedures, documentations and evaluations will be performed: descriptions of concomitant medications; hospitalisations for psychiatric reasons; clinical deterioration; Clinical Global Impression - Severity (CGI-S) and Global Assessment of Functioning (GAF) assessments; Community Treatment Order (CTO) status; weight; adherence and adverse event reporting. Physical examinations will be performed periodically. Paliperidone ER OROS will be supplied in 3 mg, 6 mg, and 9 mg tablets for oral administration. In general, the recommended Paliperidone ER dose will be 6 mg once daily, however some patients may require a higher or lower initial dose in the recommended range of 3 to 12 mg once daily. The dose can be adjusted any point during the study, to a maximum dose of 12mg/day. The study duration will be split into two phases. Phase A will be 12 weeks and Phase B which will be an optional follow up phase

ELIGIBILITY:
Inclusion Criteria:

* Patients must satisfy the following criteria to be eligible for this study: patients with diagnoses of schizophrenia according to the DSM-IV criteria including newly diagnosed patients
* Out-patients or in-patients with expected discharge within 8 weeks
* Patients or their legally acceptable representatives must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

* Patients who meet any of the following criteria will be excluded from participating in the study: patients who are resistant to antipsychotic treatment
* Patients who have been on clozapine or long-acting injectable antipsychotic medication during the last 3 months
* Patients with CGl-S scores > 6 or who who have been hospitalized for longer than 8 continuous weeks during the past 6 months
* Pregnant or breast-feeding females
* Patients with a history or current symptoms of tardive dyskinesia or neuroleptic malignant syndrome.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Pty Ltd Clinical Trial, Study Director — Janssen-Cilag Pty Ltd

REFERENCES:
- See also: An open label multicentre study to determine the dose distribution of Paliperidone ER OROS® in patients with schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=236&filename=CR013213_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Paliperidone Extended Release (ER): Paliperidone ER 3mg or 6mg or 9mg or 12mg once daily for 52 weeks
Period: Overall Study
Arm/Group | Paliperidone Extended Release (ER)
Started | 64
Completed | 32
Not Completed | 32
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 9
Not completed — Compliance | 3
Not completed — Lack of Efficacy | 3
Not completed — Adverse Event | 3
Not completed — Patient was selling medication to others | 1
Not completed — Safety evaluation | 1
Not completed — Reason not specified | 6
Not completed — Ceased in favor of Paliperidone | 1
Not completed — Switching to trial medication | 1
Not completed — No longer required | 1

BASELINE CHARACTERISTICS:
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 64
Age Continuous [Mean (Standard Deviation); unit: years] | 37.0 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: The Mean Modal Prescribed Daily Dose of Paliperidone Extended Release (ER) From Day 1 to Day 84
Time Frame: Day 1 to Day 84
Population: Intent-To-Treat (ITT) population
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 63
mg | 6.9 (2.3)

2. Primary Outcome: The Median Modal Prescribed Daily Dose of Paliperidone Extended Release (ER) From Day 1 to Day 84
Time Frame: Day 1 to Day 84
Population: Intent-To-Treat (ITT) population
Measure: Median (95% Confidence Interval); unit: mg
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 63
mg | 6 [3 to 12]

3. Primary Outcome: The Mean Modal Prescribed Daily Dose of Paliperidone Extended Release (ER) From Day 57 to Day 84
Time Frame: Day 57 to Day 84
Population: Intent-To-Treat (ITT) population, excluding participants no longer participating in the study at Day 57
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 53
mg | 7.5 (2.4)

4. Primary Outcome: The Median Modal Prescribed Daily Dose of Paliperidone Extended Release (ER) From Day 57 to Day 84
Time Frame: Day 57 to Day 84
Population: Intent-To-Treat (ITT) population, excluding participants no longer participating in the study at Day 57
Measure: Median (95% Confidence Interval); unit: mg
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 53
mg | 6 [3 to 12]

5. Primary Outcome: The Mean Overall Average Daily-prescribed Dose of Paliperidone Extended Release (ER) From Week 0 to Week 12
Time Frame: Week 0 to Week 12
Population: Intent-To-Treat (ITT) population
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 63
mg | 6.8 (1.8)

6. Primary Outcome: The Median Overall Average Daily-prescribed Dose of Paliperidone Extended Release (ER) From Week 0 to Week 12
Time Frame: Week 0 to Week 12
Population: Intent-To-Treat (ITT) population
Measure: Median (95% Confidence Interval); unit: mg
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 63
mg | 6 [3.6 to 10.3]

7. Secondary Outcome: The Clinical Global Impression of Severity (CGI-S) Throughout the Study
Description: The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a patient. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill patients".
Time Frame: 52 weeks
Population: All participants with evaluable data at each measurement time point
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Baseline; Week 2; Week 4; Week 6; Week 9; Week 12; Week 20; Week 28; Week 36; Week 44; Week 52: Paliperidone ER 3mg or 6mg or 9mg or 12mg once daily for 52 weeks
Arm/Group | Baseline | Week 2 | Week 4 | Week 6 | Week 9 | Week 12 | Week 20 | Week 28 | Week 36 | Week 44 | Week 52
Number analyzed (Participants) | 63 | 38 | 36 | 34 | 28 | 31 | 27 | 14 | 14 | 17 | 16
scores on a scale | 3.7 (1.2) | 3.3 (1.1) | 3.2 (1.0) | 3.1 (1.1) | 2.8 (1.0) | 2.8 (1.0) | 2.9 (1.1) | 2.7 (1.1) | 2.7 (0.8) | 2.9 (1.2) | 2.7 (0.8)

8. Secondary Outcome: The Global Assessment of Functioning (GAF) Throughout the Study
Description: The GAF is a 100-point tool rating overall psychological, social and occupational functioning of adults. The higher score range (91-100) refers to a superior functioning in a wide range of activities, and absence of symptoms. The lower score range (1-10) refers to persistent danger of severely hurting self or others; or persistent inability to maintain minimum personal hygiene; or serious suicidal act with clear expectation of death.
Time Frame: 52 Weeks
Population: All participants with evaluable data at each measurement time point
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Baseline | Week 2 | Week 4 | Week 6 | Week 9 | Week 12 | Week 20 | Week 28 | Week 36 | Week 44 | Week 52
Number analyzed (Participants) | 63 | 38 | 36 | 34 | 28 | 31 | 27 | 14 | 14 | 17 | 16
scores on a scale | 54.6 (14.7) | 58.9 (15.0) | 63.9 (15.3) | 63.9 (15.6) | 66.3 (13.8) | 65.4 (14.6) | 65.1 (14.7) | 71.1 (13.3) | 71.6 (14.9) | 69.0 (17.2) | 63.3 (15.7)

9. Secondary Outcome: The Percentage of Participants Presenting Clinical Deterioration Throughout the Study
Description: This Outcome Measure is intended to document only the hospitalizations associated with clinical deterioration, ie, when the patient needs to be hospitalized due to exacerbation of psychotic symptoms.
Time Frame: 52 Weeks
Population: All participants with evaluable data at each measurement time point
Measure: Number; unit: percentage of participants
Arm/Group | Baseline | Week 2 | Week 4 | Week 6 | Week 9 | Week 12 | Week 20 | Week 28 | Week 36 | Week 44 | Week 52
Number analyzed (Participants) | 63 | 38 | 36 | 34 | 28 | 31 | 27 | 14 | 14 | 17 | 16
percentage of participants
  Hospitalized | 0 (14.7) | 5.3 (15.0) | 13.5 (15.3) | 5.9 (15.6) | 7.1 (13.8) | 3.2 (14.6) | 3.7 (14.7) | 0 (13.3) | 0 (14.9) | 0 (17.2) | 12.5 (15.7)
  Care Increase | 0 | 0 | 5.4 | 2.9 | 3.6 | 3.2 | 7.4 | 0 | 0 | 5.9 | 12.5
  Suicidal | 4.8 | 5.3 | 8.1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Violent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Self Injury | 0 | 0 | 0 | 0 | 0 | 3.2 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: The Number of Hospitalizations Throughout the Study
Description: This outcome measure is intended to document all hospitalizations that occurred throughout the study.
Time Frame: 52 Weeks
Population: All participants with evaluable data at each measurement time point
Measure: Number; unit: events
Arm/Group | Baseline | Week 2 | Week 4 | Week 6 | Week 9 | Week 12 | Week 20 | Week 28 | Week 36 | Week 44 | Week 52
Number analyzed (Participants) | 63 | 38 | 36 | 34 | 28 | 31 | 27 | 14 | 14 | 17 | 16
events | 15 (14.7) | 2 (15.0) | 6 (15.3) | 2 (15.6) | 3 (13.8) | 1 (14.6) | 1 (14.7) | 0 (13.3) | 0 (14.9) | 1 (17.2) | 2 (15.7)

11. Secondary Outcome: The Length of Hospitalizations Throughout the Study
Time Frame: 52 weeks
Population: Participants who were hospitalized and had evaluable data at each measurement time point
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Baseline | Week 2 | Week 4 | Week 6 | Week 9 | Week 12 | Week 20 | Week 44 | Week 52
Number analyzed (Participants) | 15 | 1 | 3 | 2 | 2 | 1 | 1 | 1 | 2
days | 12.4 (11.5) | 66 (0) | 7.3 (6.0) | 28.0 (5.7) | 179.0 (220.6) | 34 (0) | 19 (0) | 4 (0) | 20.5 (10.6)

ADVERSE EVENTS:
Arm/Group | Paliperidone Extended Release (ER)
Serious Adverse Events (participants affected / at risk) | 27/64
Other Adverse Events (participants affected / at risk) | 51/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Extended Release (ER) (N=64)
Abdominal pain (Gastrointestinal disorders) | 1
Lethargy (General disorders) | 1
Encephalitis viral (Infections and infestations) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dystonia (Nervous system disorders) | 1
Extrapyramidal disorder (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 2
Hallucination, auditory (Psychiatric disorders) | 1
Mental disorders (Psychiatric disorders) | 2
Paranoia (Psychiatric disorders) | 2
Psychotic disorder (Psychiatric disorders) | 1
Schizoaffective disorder (Psychiatric disorders) | 2
Schizophrenia (Psychiatric disorders) | 3
Schizophrenia exacerbated (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Extended Release (ER) (N=64)
Dizziness (Cardiac disorders) | 4
Nausea (Gastrointestinal disorders) | 6
Headache (Nervous system disorders) | 7
Sedation (Nervous system disorders) | 4
Tremor (Nervous system disorders) | 6
Vision blurred (Nervous system disorders) | 4
Akathisia (Psychiatric disorders) | 6
Insomnia (Psychiatric disorders) | 10
Rash (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less